CLINICAL TRIAL: NCT04501458
Title: Western Kenya Integrated COVID-19 Response Leveraging the Community Health Strategy, Youth, and Technology to Flatten the COVID-19 Curve and Improve COVID-19 Case Detection, Isolation and Management in Western Kenya
Brief Title: Western Kenya Integrated COVID-19 Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Surgical Systems Research Group (Other)
Collaborators: Wellcome Trust (Other); Tropical Institute of Community Health (Unknown)
Responsible Party: Principal Investigator, Neema Kaseje, Founding Director, Surgical Systems Research Group
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 001
Record Dates: First submitted 2020-08-05; First posted 2020-08-06 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Covid19
Keywords: youth, community health, digital tools, capacity building
MeSH Terms: conditions — COVID-19 | interventions — Community Health Workers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Functional community health units (Experimental): Community health units with active community health workers.
  Interventions: Other: Training of youth, community health assistants and community health workers.
- Non functional community health units (No Intervention): Community health units without active community health workers.
- Health facilities with oxygen capacity (Experimental): Health facility with regular oxygen capacity.
  Interventions: Other: Training clinicians in basic critical care and the management of severe COVID-19 cases
- Health facilities without oxygen capacity (No Intervention)

INTERVENTIONS:
Other: Training of youth, community health assistants and community health workers. — Training of youth, community health assistants, and community health workers in the screening, detection, contact tracing, prevention, and management of COVID-19 with concurrent maintenance of essential health services.
  Arms: Functional community health units
Other: Training clinicians in basic critical care and the management of severe COVID-19 cases — Training clinicians in basic critical care and the management of severe COVID-19 cases with concurrent maintenance of essential health services.
  Arms: Health facilities with oxygen capacity

SUMMARY:
To respond to the COVID-19 pandemic, investigators will be deploying community health workers, equipped with mobile technology, and accompanied by youth to visit households door to door to screen for symptoms of COVID-19, isolate, test, and manage suspected cases of COVID-19. The community health workers and youth will educate households about preventive measures including frequent handwashing and home management of mild cases. Simultaneously, investigators will work with nurses, doctors, and clinical officers, to test and treat more severe cases of COVID-19 in health facilities. Our goals are: to visit every household in Siaya county covering a population of close to 1 million, and to train and support health workers working in 32 health facilities with oxygen capacity in Siaya to reduce the morbidity and mortality related to COVID19 and other conditions.

ELIGIBILITY:
Inclusion Criteria:

* Youth aged 18 to 30 years old.
* Active community health workers.
* Facilities with oxygen capacity.

Exclusion Criteria:

* Individuals younger than 18 or older than 30 years old.
* Inactive community health workers.
* Facilities without oxygen capacity.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200000 (Estimated)
Dates: Start 2020-08-10 (Actual); Primary Completion 2022-06-10 (Estimated); Study Completion 2022-06-10 (Estimated)

PRIMARY OUTCOMES:
Mortality | 3 months
  Mortality related to COVID-19
Number of confirmed COVID-19 cases in Siaya | 3 months
  Number of confirmed COVID-19 cases in Siaya

CONTACTS AND LOCATIONS:
Overall Officials: Neema Kaseje, MD, Principal Investigator — Surgical Systems Research Group
Locations (1):
- Surgical Systems Research Group/Tropical Institute of Community Health, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be available when results are reported.
Supporting Information: Study Protocol
Time Frame: Immediately following publication; indefinitely.
Access Criteria: Anyone with an approved proposal who wishes to access the data.

REFERENCES:
- See also: Full protocol — https://wellcomeopenresearch.org/articles/6-15/v1